CLINICAL TRIAL: NCT04497844
Title: A Phase 3 Randomized, Placebo-controlled, Double-blind Study of Niraparib in Combination With Abiraterone Acetate and Prednisone Versus Abiraterone Acetate and Prednisone for the Treatment of Participants With Deleterious Germline or Somatic Homologous Recombination Repair (HRR) Gene-Mutated Metastatic Castration-Sensitive Prostate Cancer (mCSPC)
Brief Title: A Study of Niraparib in Combination With Abiraterone Acetate and Prednisone Versus Abiraterone Acetate and Prednisone for the Treatment of Participants With Deleterious Germline or Somatic Homologous Recombination Repair (HRR) Gene-Mutated Metastatic Castration-Sensitive Prostate Cancer (mCSPC)
Acronym: AMPLITUDE
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR108852; 67652000PCR3002 (Other: Janssen Research & Development, LLC); 2020-002209-25 (EudraCT Number); 2023-506365-64-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2020-07-31; First posted 2020-08-04 (Actual); Results first posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Castration-sensitive Prostate Cancer
MeSH Terms: interventions — niraparib; Abiraterone Acetate; Prednisone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Niraparib with Abiraterone Acetate plus Prednisone (AAP) (Experimental): Participants will receive the following in each 28-day treatment cycle: niraparib 200 milligrams (mg), abiraterone acetate (AA) 1000 mg plus prednisone 5 mg once daily.
  Interventions: Drug: Niraparib; Drug: Abiraterone acetate (AA); Drug: Prednisone
- AA plus Prednisone (AAP) (Active Comparator): Participants will receive the following in each 28-day treatment cycle: matching placebo for Niraparib along with AA 1000 mg plus prednisone 5 mg once daily.
  Interventions: Drug: Abiraterone acetate (AA); Drug: Prednisone; Drug: Placebo for Niraparib

INTERVENTIONS:
Drug: Niraparib — Participants will receive Niraparib 200 mg once daily.
  Arms: Niraparib with Abiraterone Acetate plus Prednisone (AAP)
Drug: Abiraterone acetate (AA) — Participants will receive AA 1000 mg once daily.
Drug: Prednisone — Participants will receive prednisone 5 mg once daily.
Drug: Placebo for Niraparib — Participants will receive matching placebo for Niraparib once daily.
  Arms: AA plus Prednisone (AAP)

SUMMARY:
The purpose of the study is to determine if the combination of niraparib with Abiraterone Acetate (AA) plus prednisone compared with AA plus prednisone in participants with deleterious germline or somatic Homologous Recombination Repair (HRR) gene-mutated Metastatic Castration-Sensitive Prostate Cancer (mCSPC) provides superior efficacy in improving radiographic progression-free survival (rPFS).

DETAILED DESCRIPTION:
Prostate cancer is a heterogenous disease and recent genomic analyses have highlighted specific germline and somatic mutations and alternative driver growth signaling pathways in patients with metastatic disease. Abiraterone acetate plus prednisone (AAP) is an established standard of care for the treatment of participants with mCSPC and is included in widely accepted clinical treatment guidelines. Niraparib in combination with AAP has been approved for the treatment of BRCA-mutated Metastatic Castration-Resistant Prostate Cancer (mCRPC). Niraparib is an investigational agent in the Metastatic Castration-Sensitive Prostate Cancer (mCSPC) population. Whether the addition of niraparib to the AAP standard of care may improve initial disease control and long-term outcomes compared with AAP alone in a biomarker selected mCSPC population is being evaluated on this trial. The study will consist of 4 phases; a Prescreening Phase for biomarker evaluation for eligibility only, a Screening Phase, a Treatment Phase, and a Follow-up Phase. Efficacy evaluations include the following: tumor measurements by computed tomography (CT), magnetic resonance imaging (MRI; abdomen, chest, and pelvis), Technetium-99m (99mTc) bone scans, serum prostate sensitive antigen (PSA) evaluations, and patient reported outcomes (PROs). Safety evaluations include incidence of adverse events and clinical laboratory parameters.

ELIGIBILITY:
Inclusion criteria:

* Pathological diagnosis of prostate adenocarcinoma
* Must have appropriate deleterious homologous recombination repair (HRR) gene alteration
* Metastatic disease as documented by conventional imaging with computed tomography (CT) or magnetic resonance imaging (MRI) (for soft tissue lesions) or 99mTc bone scan (for bone lesions). Participants with a single bone lesion on Technetium-99m (99mTc) bone scan with no other non-nodal metastatic disease must have confirmation of bone metastasis by CT or MRI. Participants with lymph node-only disease are not eligible
* Androgen deprivation therapy (either medical or surgical castration) must have been started >=14 days prior to randomization and participants be willing to continue androgen deprivation therapy (ADT) through the treatment phase
* Other allowed prior therapy for metastatic castration-sensitive prostate cancer (mCSPC): (a) maximum of 1 course of radiation and 1 surgical intervention for symptomatic control of prostate cancer (example, uncontrolled pain, impending spinal cord compression or obstructive symptoms). Participants with radiation or surgical interventions to all known sites of metastatic disease will be excluded from trial participation. Radiation must be completed prior to randomization (b) Up to a maximum of 6 months of ADT prior to randomization; (c) Up to a maximum of 45 days of abiraterone acetate + prednisone (AA-P) prior to randomization (d) Up to a maximum of 2 weeks of ketoconazole for prostate cancer prior to randomization

Exclusion criteria:

* Prior treatment with a poly (adenosine diphosphate-ribose) polymerase inhibitor (PARP inhibitor)
* History of adrenal dysfunction
* Long-term use of systemically administered corticosteroids (greater than [>] 5 milligrams [mg] of prednisone or the equivalent) during the study is not allowed. Short-term use (<=4 weeks, including taper) and locally administered steroids (for example, inhaled, topical, ophthalmic, and intra-articular) are allowed, if clinically indicated
* History or current diagnosis of myelodysplastic syndrome (MDS)/ acute myeloid leukemia (AML)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 696 (Actual)
Dates: Start 2020-09-23 (Actual); Primary Completion 2025-01-07 (Actual); Study Completion 2027-11-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (387):
- United States (53):
  - Urology Centers Of Alabama, Homewood, Alabama
  - Mayo Clinic Arizona, Phoenix, Arizona
  - Urological Associates of Southern Arizona, P.C., Tucson, Arizona
  - Greater Los Angeles VA Healthcare System, Los Angeles, California
  - University of California Irvine Medical Center Chao Family Comprehensive Cancer Center, Orange, California
  - San Bernardino Urological Associates, San Bernardino, California
  - University of San Francisco California, San Francisco, California
  - Rocky Mountain Cancer Centers, Colorado Springs, Colorado
  - AdventHealth Medical Group Urology of Denver, Denver, Colorado
  - Colorado Clinical Research, Lakewood, Colorado
  - Eastern Connecticut Hematology & Oncology Assoc., Norwich, Connecticut
  - Advanced Urology Institute, Daytona Beach, Florida
  - Holy Cross Hospital - Michael and Dianne Bienes Comprehensive Cancer Center, Fort Lauderdale, Florida
  - University of Florida Health Jacksonville, Jacksonville, Florida
  - Cancer Specialists of North Florida, Jacksonville, Florida
  - Urology of Indiana, Greenwood, Indiana
  - First Urology, Jeffersonville, Indiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Baltimore VA Medical Center, Baltimore, Maryland
  - Maryland Oncology Hematology, PA, Columbia, Maryland
  - Chesapeake Urology Associates, Towson, Maryland
  - Michigan Institute of Urology, Troy, Michigan
  - Mosaic Life Care, Saint Joseph, Missouri
  - St. Louis VA Medical Center, St Louis, Missouri
  - GU Research Network, Omaha, Nebraska
  - New York Oncology Hematology, Albany, New York
  - Manhattan VAMC, New York, New York
  - Mount Sinai, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Associated Medical Professionals, Syracuse, New York
  - Montefiore Medical Center, The Bronx, New York
  - Durham VAMC, Durham, North Carolina
  - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - VA Portland Health Care System, Portland, Oregon
  - Oregon Oncology Specialists, Salem, Oregon
  - Keystone Urology Specialists, Lancaster, Pennsylvania
  - Philadelphia VA Medical Center, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center (UPMC), Pittsburgh, Pennsylvania
  - Ralph H. Johnson Veterans Affairs Medical Center, Charleston, South Carolina
  - Prisma Health, Seneca, South Carolina
  - Urology Associates, Nashville, Tennessee
  - Texas Oncology-Austin, Austin, Texas
  - Texas Oncology - Northeast, Denton, Texas
  - Houston Metro Urology, Houston, Texas
  - Texas Oncology P A, New Braunfels, Texas
  - Texas Oncology - Northeast, Tyler, Texas
  - University of Utah Huntsman Cancer Institute, Salt Lake City, Utah
  - Virginia Oncology Associates, Norfolk, Virginia
  - Virginia Commonwealth University - Massey Cancer Center, Richmond, Virginia
  - VA Puget Sound Healthcare System, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - MultiCare Health System, Tacoma, Washington
- Argentina (15):
  - Sociedade Beneficente de Senhoras Hospital Sirio Libanes, Buenos Aires
  - Centro Oncológico Korben, Buenos Aires
  - Hospital Militar Cosme Argerich, C.a.b.a.
  - CINME Centro de Investigaciones Metabolicas, Caba
  - CIPREC Arenales, CABA
  - Centro de Urologia (CDU), Ciudad Automoma Buenos Aires
  - Hospital Italiano de Buenos Aires, Ciudad Autonoma de
  - Clinica Adventista Belgrano, Ciudad de Buenos Aires
  - Cemaic Centro Privado de Especialidades Medicas Ambulatorias e Investigacion Clinica, Córdoba
  - Centro Urologico Profesor Bengio, Córdoba
  - Instituto Médico de Río Cuarto, Córdoba
  - Hospital Privado de Cordoba, Córdoba
  - Hospital Privado de Comunidad, Mar del Plata
  - Centro de Investigacion Pergamino SA, Pergamino
  - ARS Médica, San Salvador de Jujuy
- Australia (11):
  - Sunshine Coast University Hospital, Birtinya
  - St Vincent s Hospital Sydney, Darlinghurst
  - Cancer Care Services Clinical Research Unit, Herston
  - Royal Hobart Hospital, Hobart
  - Icon Cancer Centre Kurralta Park, Kurralta Park
  - Liverpool Hospital, Liverpool
  - Peter MacCallum Cancer Centre, Melbourne
  - Fiona Stanley Hospital, Murdoch
  - Macquarie University Hospital, North Ryde
  - ICON Cancer Care, South Brisbane
  - St John of God Subiaco Hospital, Subiaco
- Belarus (8):
  - Bobruisk Interregional Oncology Dispensary, Babruysk
  - Brest Regional Oncology Dispensary, Brest
  - Grodno University Hospital, Grodno
  - Gomel Regional Clinical Oncology Dispensary, Homyel
  - N N Alexandrov National Cancer Centre of Belarus, Lesnoy
  - Minsk city Clinical Oncological Dispensary, Minsk
  - Mogilev Regional Oncology Dispensary, Mogilev
  - Vitebsk Regional Clinical Oncology Dispensary, Vitebsk
- Belgium (8):
  - ZNA Middelheim, Antwerp
  - Grand Hopital De Charleroi Site Les Viviers, Charleroi
  - Jolimont, Haine-St-Paul
  - CHC MontLegia, Liège
  - CHU UCL Namur - Site Sainte Elisabeth, Namur
  - Clinique St Pierre, Ottignies
  - Algemeen Ziekenhuis Delta, Roeselare
  - GZA Ziekenhuizen, Wilrijk
- Brazil (31):
  - Fundacao Pio XII, Barretos
  - Cetus Oncologia, Belo Horizonte
  - PERSONAL Oncologia de Precisao e Personalizada, Belo Horizonte
  - CIONC Centro Integrado de Oncologia de Curitiba, Curitiba
  - Centro de Pesquisa e Ensino em Oncologia de Santa Catarina CEPEN, Florianópolis
  - Pronutrir, Fortaleza
  - Associacao de Combate ao Cancer em Goias - Hospital de Cancer Araujo Jorge, Goiânia
  - Fundacao Sao Francisco Xavier, Ipatinga
  - Instituto Joinvilense de Hematologia e Oncologia Ltda Centro de Hematologia e Oncologia, Joinville
  - Liga Norte Riograndense Contra O Cancer, Natal
  - UPCO Unidade de Pesquisa Clinica em Oncologia, Pelotas
  - Irmandade Santa Casa de Misericordia de Porto Alegre, Porto Alegre
  - Hospital Ernesto Dornelles, Porto Alegre
  - MultiHemo Servicos Medicos S.A, Recife
  - Ministerio da Saude Instituto Nacional do Cancer, Rio de Janeiro
  - Universidade do Estado do Rio de Janeiro - UERJ, Rio de Janeiro
  - Oncoclinicas Rio de Janeiro S A, Rio de Janeiro
  - Instituto de Educacao, Pesquisa e Gestao em Saude Instituto Americas (COI), Rio de Janeiro
  - Nucleo de Oncologia da Bahia, Salvador
  - Hospital Sao Rafael, Salvador
  - Fundacao do ABC Centro Universitario FMABC, Santo André
  - Instituto do Cancer Arnaldo Vieira de Carvalho, São Paulo
  - Irmandade Santa Casa de Misericordia de Sao Paulo, São Paulo
  - Instituto de Ensino e Pesquisa São Lucas, São Paulo
  - Fundacao Faculdade de Medicina - Instituto do Cancer do Estado de Sao Paulo, São Paulo
  - Real e Benemerita Associacao Portuguesa de Beneficencia, São Paulo
  - Hospital Alemao Oswaldo Cruz, São Paulo
  - Núcleo de Pesquisa São Camilo, São Paulo
  - Instituto de Assistencia Medica ao Servidor Publico Estadual IAMSPE, São Paulo
  - IOS - Instituto de Oncologia de Sorocaba Dr. Gilson Delgado, Sorocaba
  - Centro Oncológico do Triângulo, Uberlândia
- Bulgaria (7):
  - MHAT Deva Maria, Burgas
  - UMHAT 'Dr. Georgi Stranski', EAD, Pleven
  - Complex Oncology Center - Plovdiv EOOD, Plovdiv
  - Multifunctional Hospital for Active Treatment for Women Health Nadezhda, Sofia
  - Specialized Hospital for Active Treatment in Oncology, Sofia
  - UMHAT Sofia Med, Sofia
  - Comprehensive Cancer Center, Vratsa
- Canada (11):
  - Prostate Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - British Columbia Cancer Agency(BCCA)-Sindi Ahluwalia Hawkins Centre for the Southern Interior(CSI), Kelowna, British Columbia
  - British Columbia Cancer Agency BCCA Vancouver Centre, Vancouver, British Columbia
  - British Columbia Cancer Agency Vancouver Island Centre, Victoria, British Columbia
  - McMaster Institute of Urology, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston General Health Research Institute, Kingston, Ontario
  - Sunnybrook Health Sciences Center, Toronto, Ontario
  - Princess Margaret Cancer Centre University Health Network, Toronto, Ontario
  - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - McGill University - Jewish General Hospital, Montreal, Quebec
- China (30):
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing
  - Peking University First Hospital, Beijing
  - Beijing Friendship Hospital Capital Medical University, Beijing
  - Beijing Cancer Hospital, Beijing
  - Beijing University Third Hospital, Beijing
  - Beijing Hospital, Beijing
  - West China Hospital of Sichuan University, Chengdu
  - Sichuan Provincial Peoples Hospital, Chengdu
  - Western Theater General Hospital of the Chinese People's Liberation Army, Chengdu
  - Chongqing University Cancer Hospital, Chongqing
  - Southwest Hospital, The Third Military Medical University, Chongqing
  - Sun Yat Sen University Cancer Center, Guangzhou
  - Guangzhou First Municipal People's Hospital, Guangzhou
  - Sun Yat-Sen Memorial Hospital, Sun Yat-Sen University, Guangzhou
  - Zhejiang Provincial People's Hospital, Hangzhou
  - The First Affiliated Hospital of NanChang University, Nanchang
  - Jiangsu Province Cancer Hospital, Nanjing
  - Nanjing Drum Tower Hospital, Nanjing
  - The First Affiliated Hospital of Ningbo University, Ningbo
  - Fudan University Shanghai Cancer Center, Shanghai
  - Huashan Hospital Fudan University, Shanghai
  - Renji Hospital Affiliated to Medical College of Shanghai Jiaotong University, Shanghai
  - The Fifth People's Hospital of Shanghai, Fudan University, Shanghai
  - Huadong Hospital Affiliated to Fudan University, Shanghai
  - Shengjing Hospital Of China Medical University, Shenyang
  - Second Affiliated Hospital of Soochow University, Suzhou
  - The First Affliated Hospital of Soochow University, Suzhou
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou
  - TongJi Hospital of TongJi Medical College of Huazhong University of Science & Technology, Wuhan
  - The First Affiliated Hospital of Xian Jiaotong University, Xi'an
- Czechia (5):
  - Fakultni nemocnice u sv. Anny v Brne, Brno
  - FN Hradec Kralove, Urologicka klinika, Hradec Králové
  - Krajská nemocnice Liberec, Liberec
  - Uromedical Center s.r.o., Olomouc
  - Urologicka klinika 1 LF UK a VFN, Prague
- Denmark (6):
  - Aalborg University Hospital, Aalborg
  - Copenhagen University Hospital, Copenhagen
  - Herlev Hospital, Herlev
  - Næstved Hospital, Næstved
  - Odense Universitetshospital, Odense
  - Vejle Hospital, Vejle
- France (18):
  - Institut de Cancerologie de l Ouest ICO, Angers
  - Institut Sainte Catherine, Avignon
  - CHRU De Besancon, Besançon
  - Institut Bergonie, Bordeaux
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Georges Francois Leclerc, Dijon
  - Centre Oscar Lambret, Lille
  - Centre Leon Berard, Lyon
  - Hopital Prive Jean Mermoz, Lyon
  - Institut Regional du Cancer de Montpellier Val d'Aurelle, Montpellier
  - Polyclinique de Gentilly, Nancy
  - CHU De Poitiers, Poitiers
  - Centre Hopitalier Inter-Communal De Cornouaille, Quimper
  - HIA Begin, Saint-Mandé
  - Institut de Cancérologie de Loire, Saint-Priest-en-Jarez
  - Clinique Sainte Anne, Strasbourg
  - Hopital Foch, Suresnes
  - CHRU de Tours, Tours
- Germany (8):
  - Städtisches Klinikum Braunschweig gGmbH - Standort Salzdahlumer, Braunschweig
  - Universitaetsklinikum Koelnt, Cologne
  - Universitätsklinik Carl Gustav Carus, Med. Klinik u. Poliklinik I, Dresden
  - Urologicum Duisburg, Duisburg
  - Medizinische Hochschule Hannover, Hanover
  - Klinikum rechts der Isar - III. Med. Klinik und Poliklinik, München
  - Universitaetsklinikum Muenster, Münster
  - Studienpraxis Urologie Drs. Feyerabend, Nürtingen
- Hungary (7):
  - Jahn Ferenc Del-pesti Korhaz es Rendelointezet, Budapest
  - Debreceni Egyetem, Debrecen
  - Petz Aladar Megyei Oktato Korhaz, Győr
  - Bekes Megyei Kozponti Korhaz Pandy Kalman Tagkorhaz, Gyula
  - Borsod Abauj Zemplen Varmegyei Kozponti Korhaz es Egyetemi Oktato Korhaz, Miskolc
  - Szegedi Tudomanyegyetem, Szeged
  - Szent Borbala Hospital Tatabanya, Tatabánya
- Israel (7):
  - Haemek Medical Center - Afula, Afula
  - Soroka Hospital, Beersheba
  - Rambam Medical Center, Haifa
  - Hadassah Hospital, Jerusalem
  - Rabin Medical Center, Beilinson Hospital, Petach Tikvah
  - Sheba Medical Center Tel Hashomer, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (16):
  - Ospedale S. Donato - Asl 8 Arezzo, Arezzo
  - Divisione di Oncologia - Istituto per la ricerca e cura del cancro, Candiolo
  - Istituti Ospitalieri di Cremona, AO di Cremona, Cremona
  - Azienda Ospedaliera ''Vito Fazzi'', Lecce
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori, Meldola
  - Ospedale San Raffaele, Milan
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - European Institute of Oncology, Milan
  - Fondazione G Pascale Istituto Nazionale Tumori IRCCS, Napoli
  - Aou San Luigi Gonzaga, Orbassano
  - Istituto Oncologico Veneto Iov Irccs Padova, Padua
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - ASL Napoli 2 Nord-SM delle Grazie Hospital, Pozzuoli
  - Casa Sollievo Della Sofferenza IRCCS, San Giovanni Rotondo
  - Ospedale S. Chiara, Trento
  - Ospedale San Bortolo, Vicenza
- Malaysia (6):
  - Hospital Pulau Pinang, George Town
  - Hospital Sultan Ismail, Johor Bahru
  - Hospital Kuala Lumpur, Kuala Lumpur
  - University Malaya Medical Centre, Kuala Lumpur
  - Sarawak General Hospital, Kuching
  - Institut Kanser Negara Clinical Research Center, Putrajaya
- Mexico (8):
  - Consultorio de Especialidad en Urologia Privado, Durango
  - Consultorio Privado, León
  - Centro de Investigación Clínica Gramel S.C., Mexico City
  - Avix Investigacion Clinica S C, Monterrey
  - i Can Oncology Center, Monterrey
  - Oncologia Integral Satelite, Naucalpan
  - Centro de Investigacion Clinica de Oaxaca, Oaxaca City
  - Consultorio Privado, Zapopan
- Netherlands (4):
  - Reinier de Graaf Gasthuis, Delft
  - Tergooiziekenhuizen, Hilversum
  - Canisius-Wilhelminaziekenhuis, Nijmegen
  - Elisabeth-TweeSteden Ziekenhuis, Tilburg
- New Zealand (4):
  - Auckland City Hospital, Auckland
  - Canterbury Urology Research Trust, Christchurch
  - Dunedin Hospital, Dunedin Central
  - Tauranga Hospital, Tauranga
- Poland (11):
  - IN VIVO Sp. z o.o, Bydgoszcz
  - Szpital Uniwersytecki NR 1 IM Dr Antoniego Jurasza, Bydgoszcz
  - Centrum Onkologii im Prof F Lukaszczyka, Bydgoszcz
  - Szpitale Pomorskie Sp z o o, Gdynia
  - Przychodnia Lekarska KOMED Roman Karaszewski, Konin
  - Klinika MedTrials, Krakow
  - Wojewodzki Szpital Specjalistyczny im. M. Kopernika w Lodzi, Lodz
  - Medisport, Lublin
  - Urologica Praktyka Lekarska Adam Marcheluk, Siedlce
  - Szpital Grochowski Im Dr Med Rafala Masztaka Sp Z O O, Warsaw
  - Specjalistyczna przychodnia lekarska POLIMED, Wroclaw
- Portugal (4):
  - Uls Almada Seixal - Hosp. Garcia de Orta, Almada
  - Instituto Português de Oncologia Francisco Gentil - Centro Regional de Oncologia de Coimbra, S.A., Coimbra
  - Fund. Champalimaud, Lisbon
  - Uls Santa Maria - Hosp. Santa Maria, Lisbon
- Puerto Rico Medical Research Center, Hato Rey, Puerto Rico
- Russia (15):
  - Altai Regional Oncology Dispensary, Barnaul
  - Chelyabinsk Regional Clinical Center Of Oncology And Nuclear Medicine, Chelyabinsk
  - Ivanovo Regional Oncology Dispensary, Ivanovo
  - Moscow City Clinical Hospital # 62, Moscow
  - Hertzen Oncology Research Institute, Moscow
  - Privolzhsky District Medical Centre, Nizhny Novgorod
  - Clinical Oncology Dispensary, Omsk
  - LLC Novaya Clinica, Pyatigorsk
  - Pyatigorsk Interdistrict Oncology Dispensary, Pyatigorsk
  - Leningrad Regional Oncology Dispensary, Saint Petersburg
  - Private Medical Institution Euromedservice, Saint Petersburg
  - Republican Oncology Dispensary, Saransk
  - Tomsk Cancer Research Institute, Tomsk
  - Multifunctional clinical medical center 'Medical city', Tyumen
  - Bashkir State Medical University, Ufa
- South Africa (3):
  - CancerCare Rondebosch, Cape Town
  - Steve Biko Academic Hospital, Pretoria
  - East Rand Urology Research Unit, Vosloorus
- South Korea (14):
  - Pusan National University Hospital, Busan
  - Kyungpook National University Chilgok Hospital, Daegu
  - Keimyung University Dongsan Hospital, Daegu
  - Chungnam National University Hospital, Daejeon
  - Chonnam National University Hospital, Gwangju
  - National Cancer Center, Gyeonggi-do
  - Ajou University Hospital, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si
  - Seoul National University Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital, Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea Seoul St Mary s Hospital, Seoul
- Spain (16):
  - Hosp Univ A Coruna, A Coruña
  - Hosp. de La Santa Creu I Sant Pau, Barcelona
  - Hosp Clinic de Barcelona, Barcelona
  - Hosp. Gral. Univ. de Castellon, Castellon
  - Institut Català D'Oncologia Girona, Girona
  - Hosp. de Jerez de La Frontera, Jerez de la Frontera
  - Hosp. Univ. de La Princesa, Madrid
  - Hosp. Univ. Ramon Y Cajal, Madrid
  - Hosp. Univ. 12 de Octubre, Madrid
  - Hosp. Univ. La Paz, Madrid
  - Hosp. Univ. Hm Monteprincipe, Madrid
  - Hosp Virgen de La Victoria, Málaga
  - Corporacio Sanitari Parc Tauli, Sabadell
  - Hosp. Univ. Marques de Valdecilla, Santander
  - Hosp. Virgen Del Rocio, Seville
  - Hosp. Clinico Univ. de Valencia, Valencia
- Sweden (4):
  - Salgrenska University hospital, Gothenburg
  - Urologiska Mottagningen, Malmo
  - Sodersjukhuset, Stockholm
  - Karolinska Universitetssjukhuset Solna, Stockholm
- Taiwan (8):
  - Kaohsiung Medical University Chung Ho Memorial Hospital, Kaohsiung City
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - Tungs' Taichung MetroHarbor Hospital, Taichung
  - National Taiwan University Hospital., Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang-Gung Memorial Hospital, LinKou Branch, Taoyuan District
- Thailand (3):
  - King Chulalongkorn Memorial Hospital, Bangkok
  - Ramathibodi Hospital, Bangkok
  - Siriraj Hospital, Bangkok
- Turkey (Türkiye) (16):
  - Adana Baskent Yuregir Hospital, Adana
  - Dr Abdurrahman Yurtaslan Oncology Training and Research Hospital, Ankara
  - Memorial Ankara Hastanesi, Ankara
  - Gazi University Hospital, Ankara
  - Ankara University Medical Faculty, Ankara
  - Ankara Bilkent City Hospital, Ankara
  - Bursa Yuksek lhtisas EAH Medikal Onkoloji Klinigi, Bursa
  - Trakya University Medical Faculty, Edirne
  - Istanbul University Istanbul Medical Faculty, Istanbul
  - Istanbul Universitesi Cerrahpasa Tip Fakultesi Ic Hastaliklari Anabilim Dali Medikal Onkoloji Bd, Istanbul
  - Bakirkoy Training and Research Hospital, Istanbul
  - T C Saglik Bakanlıgi Goztepe Prof Dr Suleyman Yalcın Sehir Hastanesi, Istanbul
  - Dokuz Eylul University Medical Faculty, Izmir
  - Izmir Medical Point Hospital, Izmir
  - Sakarya University Training and Research Hospital, Sakarya
  - Medical Park Samsun Hastanesi, Samsun
- Ukraine (16):
  - CNE Clinical Center of Oncology Hematology Transplantology and Palliative Care of the Cherkasy RC, Cherkasy
  - Municipal Non-profit enterprise 'Bukovinian clinical oncology center', Chernivtsi
  - Ce 'Dnipropetrovsk Regional Clinical Hospital N.A. Mechnikov' of Dnipropetrovsk Rc, Dnipro
  - Municipal Institution 'Clinical Oncology Dispensary' Under Dnipropetrovsk Regional Council, Dnipro
  - Dnipropetrovsk State Medical Academy, Dnipropetrovsk City Multifield Clinical Hospital # 4, Dnipro
  - Ivano-Frankivsk Regional Clinical Hospital, Ivano-Frankivsk
  - Communal Institution 'City hospital №7 of Kamianske' of Dnepropetrov'sk Regional Council, Kamianske
  - Municipal non-profit enterprise 'Regional Center of Oncology', Khakhiv
  - Regional Medical Clinical Center for Urology and Nephrology named after V.I. Shapoval, Kharkiv
  - Kherson Regional Oncological Dispensary, Kherson
  - Nonprofit Organization National Cancer Institute, Kyiv
  - State Institution Institute of Urology NAMS of Ukraine based on Kyiv City Clinical Oncology Center, Kyiv
  - Kyiv Regional Oncological Dispensary, Kyiv
  - Communal Noncommercial Enterprise of Lviv Regional Council 'Lviv Regional Clinical Hospital', Lviv
  - Podilskiy Regional Center of Oncology, Vinnitsa
  - Communal Institution 'Regional Oncology Dispensary' of Zhytomyr Region Council, Zhytomyr
- United Kingdom (13):
  - Ysbyty Gwynedd, Bangor
  - Belfast City Hospital, Belfast
  - Brighton and Sussex University Hospitals NHS Trust, Brighton
  - Bristol Haematology and Oncology Centre, Bristol
  - Guy's Hospital, Great Maze Pond
  - Prince Of Wales Hospital, Grimsby
  - Marie Curie Research Wing - Mount Vernon Hospital, Hillingdon
  - Raigmore Hospital, Inverness
  - University College London Hospitals NHSFT, London
  - Churchill Hospital, Oxford
  - Royal Preston Hospital, Preston
  - Royal Marsden Hospital, Sutton
  - Royal Cornwall Hospitals NHS Trust - Royal Cornwall Hospital, Truro

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] Attard G, Agarwal N, Graff JN, Sandhu S, Efstathiou E, Ozguroglu M, Pereira de Santana Gomes AJ, Vianna K, Luo H, Gotto GT, Cheng HH, Kim W, Varela CR, Schaeffer D, Kramer K, Li S, Baron B, Shen F, Mundle SD, McCarthy SA, Olmos D, Chi KN, Rathkopf DE. Niraparib and abiraterone acetate plus prednisone for HRR-deficient metastatic castration-sensitive prostate cancer: a randomized phase 3 trial. Nat Med. 2025 Dec;31(12):4109-4118. doi: 10.1038/s41591-025-03961-8. Epub 2025 Oct 7. PMID 41057655

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The results presented are based on the primary completion date (07 January 2025). Remaining results will be reported within a year of study completion.
Groups:
- Placebo With Abiraterone Acetate Plus Prednisone: Participants with deleterious germline or somatic homologous recombination repair (HRR) gene-mutated metastatic castration- sensitive prostate cancer (mCSPC) were randomized to receive placebo matching to niraparib and abiraterone acetate (AA) fixed dose combination (FDC) tablets along with AA tablets (4*250 mg tablet) and prednisone 5 mg tablet orally, once daily from Day 1 of Cycle 1 up to 49 cycles. Each treatment cycle consisted of 28 days.
- Niraparib With Abiraterone Acetate Plus Prednisone: Participants with deleterious germline or somatic HRR gene-mutated mCSPC were randomized to receive niraparib and AA FDC tablets (2* [100 mg niraparib/500 mg AA tablet]) along with placebo matching to AA tablet and prednisone 5 mg tablet orally, once daily from Day 1 of Cycle 1 up to 49 cycles. Each treatment cycle consisted of 28 days.
Period: Overall Study
Arm/Group | Placebo With Abiraterone Acetate Plus Prednisone | Niraparib With Abiraterone Acetate Plus Prednisone
Started | 348 | 348
Treated | 348 | 347
BRCA Subgroup | 196 | 191
HRR Effector Subgroup | 226 | 230
All HRR | 348 | 348
Completed | 0 | 0
Not Completed | 348 | 348
Not completed — Ongoing | 231 | 249
Not completed — Death | 106 | 84
Not completed — Lost to Follow-up | 2 | 0
Not completed — Withdrawal by Subject | 6 | 14
Not completed — Regional Crisis | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo With Abiraterone Acetate Plus Prednisone | Niraparib With Abiraterone Acetate Plus Prednisone | Total
Number analyzed (Participants) | 348 | 348 | 696
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.7 (8.84) | 67.8 (8.75) | 67.3 (8.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 348 | 348 | 696
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 43 | 40 | 83
  Not Hispanic or Latino | 292 | 287 | 579
  Unknown or Not Reported | 13 | 21 | 34
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 1 | 4
  Asian | 67 | 77 | 144
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 10 | 18 | 28
  White | 257 | 246 | 503
  More than one race | 2 | 2 | 4
  Unknown or Not Reported | 8 | 4 | 12
Age, Categorical [Count of Participants; unit: Participants]
  Adults (18-64 years) | 135 | 116 | 251
  From 65 to 84 years | 212 | 227 | 439
  85 years and over | 1 | 5 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  ARGENTINA | 15 | 15 | 30
  AUSTRALIA | 9 | 14 | 23
  BELARUS | 6 | 1 | 7
  BELGIUM | 4 | 5 | 9
  BRAZIL | 30 | 28 | 58
  BULGARIA | 3 | 2 | 5
  CANADA | 14 | 15 | 29
  CHINA | 24 | 29 | 53
  CZECH REPUBLIC | 3 | 3 | 6
  DENMARK | 6 | 4 | 10
  FRANCE | 17 | 15 | 32
  GERMANY | 6 | 6 | 12
  HUNGARY | 4 | 3 | 7
  ISRAEL | 3 | 11 | 14
  ITALY | 32 | 24 | 56
  MALAYSIA | 4 | 11 | 15
  MEXICO | 3 | 1 | 4
  NETHERLANDS | 2 | 1 | 3
  NEW ZEALAND | 6 | 3 | 9
  POLAND | 12 | 13 | 25
  PORTUGAL | 1 | 1 | 2
  RUSSIAN FEDERATION | 11 | 9 | 20
  SOUTH AFRICA | 1 | 2 | 3
  SOUTH KOREA | 20 | 19 | 39
  SPAIN | 18 | 21 | 39
  SWEDEN | 2 | 3 | 5
  TAIWAN | 11 | 10 | 21
  THAILAND | 4 | 3 | 7
  TURKEY | 24 | 21 | 45
  UKRAINE | 12 | 14 | 26
  UNITED KINGDOM | 11 | 11 | 22
  UNITED STATES | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Breast Cancer Gene (BRCA) Subgroup: Radiographic Progression-free Survival (rPFS) Assessed by Investigator
Description: rPFS: time interval from date of randomization to first date of radiographic progression as assessed by investigator or death due to any cause, whichever occurred first. rPFS was determined by: (1) progression of soft tissue lesions measured by computerized tomography (CT) or magnetic resonance imaging (MRI) per response evaluation criteria in solid tumors (RECIST) 1.1; (2) progression of bone lesions observed by bone scan per prostate cancer working group 3 (PCWG3) criteria: bone progression was confirmed by subsequent scan greater than or equal to (>=) 6 weeks later. Week 8 scan was baseline to which all subsequent scans were compared to determine progression. A confirmatory scan with >=2 new lesions indicated progression; A confirmatory scan not showing >=2 new lesions means no progression. If Week 8 scan shows <2 new bone lesions compared to baseline, first scan with >=2 new lesions compared to Week 8 scan indicated progression, when confirmed by a subsequent scan >=6 weeks later.
Time Frame: From date of randomization (Day -3 to Day 1) up to approximately 49 months
Population: BRCA full analysis set (FAS) included all randomized participants with BRCA gene alteration classified according to their assigned treatment arm, regardless of the actual treatment received.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- BRCA Subgroup: Placebo With Abiraterone Acetate Plus Prednisone: Participants with deleterious germline or mCSPC and BRCA alterations were randomized to receive placebo matching to niraparib and AA fixed dose combination (FDC) tablets along with AA tablets (4*250 mg tablet) and prednisone 5 mg tablet orally, once daily from Day 1 of Cycle 1 up to 49 cycles. Each treatment cycle consisted of 28 days.
- BRCA Subgroup: Niraparib With Abiraterone Acetate Plus Prednisone: Participants with deleterious germline or somatic HRR gene-mutated mCSPC and BRCA alterations were randomized to receive niraparib and AA FDC tablets (2* [100 mg niraparib/500 mg AA tablet]) along with placebo matching to AA tablet and prednisone 5 mg tablet orally, once daily from Day 1 of Cycle 1 up to 49 cycles. Each treatment cycle consisted of 28 days.
Arm/Group | BRCA Subgroup: Placebo With Abiraterone Acetate Plus Prednisone | BRCA Subgroup: Niraparib With Abiraterone Acetate Plus Prednisone
Number analyzed (Participants) | 196 | 191
months | 25.99 [22.11 to 41.17] | NA [41.20 to NA] — Median and the upper limit of the 95% confidence interval (CI) were not estimable due to an insufficient number of participants with events.
Statistical Analysis 1: Comparison: BRCA Subgroup: Placebo With Abiraterone Acetate Plus Prednisone vs BRCA Subgroup: Niraparib With Abiraterone Acetate Plus Prednisone; Test type: Superiority; p < 0.0001, Log Rank — The priori threshold for statistical significance was 0.05; Hazard Ratio (HR) = 0.515, 95% CI 2-sided [0.370 to 0.717]

2. Primary Outcome: HRR Effector Subgroup: Radiographic Progression-free Survival (rPFS) Assessed by Investigator
Description: rPFS: time interval from date of randomization to first date of radiographic progression as assessed by investigator or death due to any cause, whichever occurred first. rPFS was determined by: (1) progression of soft tissue lesions measured by CT or MRI per RECIST 1.1; (2) progression of bone lesions observed by bone scan per PCWG3 criteria: bone progression was confirmed by subsequent scan >= 6 weeks later. Week 8 scan was baseline to which all subsequent scans were compared to determine progression. A confirmatory scan with >=2 new lesions indicated progression; A confirmatory scan not showing >=2 new lesions means no progression. If Week 8 scan shows <2 new bone lesions compared to baseline, first scan with >=2 new lesions compared to Week 8 scan indicated progression, when confirmed by a subsequent scan >=6 weeks later.
Time Frame: From date of randomization (Day -3 to Day 1) up to approximately 49 months
Population: HRR effector FAS included all randomized HRR effector participants classified according to their assigned treatment arm, regardless of the actual treatment received.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- HRR Effector Subgroup: Placebo With Abiraterone Acetate Plus Prednisone: Participants with deleterious germline or gene-mutated mCSPC and HRR effector gene alterations were randomized to receive placebo matching to niraparib and AA fixed dose combination (FDC) tablets along with AA tablets (4*250 mg tablet) and prednisone 5 mg tablet orally, once daily from Day 1 of Cycle 1 up to 49 cycles. Each treatment cycle consisted of 28 days.
- HRR Effector Subgroup: Niraparib With Abiraterone Acetate Plus Prednisone: Participants with deleterious germline or somatic HRR gene-mutated mCSPC and HRR effector gene alterations were randomized to receive niraparib and AA FDC tablets (2* [100 mg niraparib/500 mg AA tablet]) along with placebo matching to AA tablet and prednisone 5 mg tablet orally, once daily from Day 1 of Cycle 1 up to 49 cycles. Each treatment cycle consisted of 28 days.
Arm/Group | HRR Effector Subgroup: Placebo With Abiraterone Acetate Plus Prednisone | HRR Effector Subgroup: Niraparib With Abiraterone Acetate Plus Prednisone
Number analyzed (Participants) | 226 | 230
months | 27.56 [25.59 to NA] — The upper limit of the 95% CI was not estimable due to an insufficient number of participants with events. | NA [41.20 to NA] — Median and the upper limit of the 95% CI were not estimable due to an insufficient number of participants with events.
Statistical Analysis 1: Comparison: HRR Effector Subgroup: Placebo With Abiraterone Acetate Plus Prednisone vs HRR Effector Subgroup: Niraparib With Abiraterone Acetate Plus Prednisone; Test type: Superiority; p = 0.0003, Log Rank — The priori threshold for statistical significance was 0.025; Hazard Ratio (HR) = 0.571, 95% CI 2-sided [0.421 to 0.774]

3. Primary Outcome: All HRR: Radiographic Progression-free Survival (rPFS) Assessed by Investigator
Description: as for outcome 2
Time Frame: From date of randomization (Day -3 to Day 1) up to approximately 49 months
Population: All HRR FAS included all randomized participants classified according to their assigned treatment arm, regardless of the actual treatment received.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo With Abiraterone Acetate Plus Prednisone | Niraparib With Abiraterone Acetate Plus Prednisone
Number analyzed (Participants) | 348 | 348
months | 29.54 [25.82 to NA] — The upper limit of the 95% CI was not estimable due to an insufficient number of participants with events. | NA [41.20 to NA] — Median and the upper limit of the 95% CI were not estimable due to an insufficient number of participants with events.
Statistical Analysis 1: Comparison: Placebo With Abiraterone Acetate Plus Prednisone vs Niraparib With Abiraterone Acetate Plus Prednisone; Test type: Superiority; p = 0.0001, Log Rank — The priori threshold for statistical significance was 0.02475; Hazard Ratio (HR) = 0.625, 95% CI 2-sided [0.490 to 0.799]

4. Secondary Outcome: BRCA Subgroup: Time to Symptomatic Progression
Description: Time to symptomatic progression was defined as time from the date of randomization to the date of any of the following (whichever occurred first): (a) the use of external beam radiation therapy for skeletal or pelvic symptoms, (b) the need for tumor-related orthopedic surgical intervention, (c) other cancer-related procedures (example: nephrostomy insertion, bladder catheter insertion, external beam radiation therapy, or surgery for tumor symptoms), (d) cancer-related morbid events (that is, fracture [symptomatic and/or pathologic], cord compression, urinary obstructive events), (e) initiation of a new systemic anti-cancer therapy because of cancer symptoms.
Time Frame: From date of randomization (Day -3 to Day 1) up to approximately 49 months
Population: BRCA FAS included all randomized participants with BRCA gene alteration classified according to their assigned treatment arm, regardless of the actual treatment received.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- BRCA Subgroup: Placebo With Abiraterone Acetate Plus Prednisone: Participants with deleterious germline or gene-mutated mCSPC and BRCA alterations were randomized to receive placebo matching to niraparib and AA fixed dose combination (FDC) tablets along with AA tablets (4*250 mg tablet) and prednisone 5 mg tablet orally, once daily from Day 1 of Cycle 1 up to 49 cycles. Each treatment cycle consisted of 28 days.
Arm/Group | BRCA Subgroup: Placebo With Abiraterone Acetate Plus Prednisone | BRCA Subgroup: Niraparib With Abiraterone Acetate Plus Prednisone
Number analyzed (Participants) | 196 | 191
months | NA [39.72 to NA] — Median and upper limit of 95% CI were not estimable due to an insufficient number of participants with events. | NA [NA to NA] — Median, lower and upper limit of 95% CI were not estimable due to an insufficient number of participants with events.
Statistical Analysis 1: Comparison: BRCA Subgroup: Placebo With Abiraterone Acetate Plus Prednisone vs BRCA Subgroup: Niraparib With Abiraterone Acetate Plus Prednisone; Test type: Superiority; p = 0.0001, Log Rank — The priori threshold for statistical significance was 0.03426; Hazard Ratio (HR) = 0.444, 95% CI 2-sided [0.290 to 0.681]

5. Secondary Outcome: HRR Effector Subgroup: Time to Symptomatic Progression
Description: as for outcome 4
Time Frame: From date of randomization (Day -3 to Day 1) up to approximately 49 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | HRR Effector Subgroup: Placebo With Abiraterone Acetate Plus Prednisone | HRR Effector Subgroup: Niraparib With Abiraterone Acetate Plus Prednisone
Number analyzed (Participants) | 226 | 230
months | NA [NA to NA] — Median, lower and upper limit of 95% CI were not estimable due to an insufficient number of participants with events. | NA [41.40 to NA] — Median and upper limit of 95% CI were not estimable due to an insufficient number of participants with events.
Statistical Analysis 1: Comparison: HRR Effector Subgroup: Placebo With Abiraterone Acetate Plus Prednisone vs HRR Effector Subgroup: Niraparib With Abiraterone Acetate Plus Prednisone; Test type: Superiority; p = 0.0004, Log Rank — The priori threshold for statistical significance was 0.02977; Hazard Ratio (HR) = 0.495, 95% CI 2-sided [0.332 to 0.738]

6. Secondary Outcome: All HRR: Time to Symptomatic Progression
Description: as for outcome 4
Time Frame: From date of randomization (Day -3 to Day 1) up to approximately 49 months
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo With Abiraterone Acetate Plus Prednisone | Niraparib With Abiraterone Acetate Plus Prednisone
Number analyzed (Participants) | 348 | 348
months | NA [43.14 to NA] — Median and upper limit of 95% CI were not estimable due to an insufficient number of participants with events. | NA [NA to NA] — Median, lower and upper limit of 95% CI were not estimable due to an insufficient number of participants with events.
Statistical Analysis 1: Comparison: Placebo With Abiraterone Acetate Plus Prednisone vs Niraparib With Abiraterone Acetate Plus Prednisone; Test type: Superiority; p < 0.0001, Log Rank — The priori threshold for statistical significance was 0.03207; Hazard Ratio (HR) = 0.503, 95% CI 2-sided [0.364 to 0.695]

7. Secondary Outcome: Overall Survival (OS)
Time Frame: From date of randomization (Day -3 to Day 1) up to 83 months
Reporting Status: Not Posted, anticipated posting 2028-11

8. Secondary Outcome: Time to Subsequent Therapy
Time Frame: From date of randomization (Day -3 to Day 1) up to 83 months
Reporting Status: Not Posted, anticipated posting 2028-11

9. Secondary Outcome: Number of Participants With Treatment-emergent Serious Adverse Events
Time Frame: From Cycle 1 Day 1 up to 83 months
Reporting Status: Not Posted, anticipated posting 2028-11

10. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events by Severity
Time Frame: From Cycle 1 Day 1 up to 83 months
Reporting Status: Not Posted, anticipated posting 2028-11

ADVERSE EVENTS:
Time Frame: All cause mortality: From screening (Day -38 up to Day -1) up to approximately 49 months. Serious adverse events (SAEs) and other AEs: From Cycle 1 Day 1 up to approximately 49 months
Description: All cause mortality: All randomized participants; SAE and Other AEs: The safety analysis set included all randomized participants who received at least 1 dose of study medication.
Arm/Group | Placebo With Abiraterone Acetate Plus Prednisone | Niraparib With Abiraterone Acetate Plus Prednisone
All-Cause Mortality (participants affected / at risk) | 108/348 | 85/348
Serious Adverse Events (participants affected / at risk) | 96/348 | 136/347
Other Adverse Events (participants affected / at risk) | 326/348 | 338/347
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo With Abiraterone Acetate Plus Prednisone (N=348) | Niraparib With Abiraterone Acetate Plus Prednisone (N=347)
Anaemia (Blood and lymphatic system disorders) | 4 | 20
Disseminated Intravascular Coagulation (Blood and lymphatic system disorders) | 0 | 1
Haemolytic Anaemia (Blood and lymphatic system disorders) | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 3
Acute Coronary Syndrome (Cardiac disorders) | 0 | 1
Acute Myocardial Infarction (Cardiac disorders) | 3 | 0
Angina Pectoris (Cardiac disorders) | 3 | 0
Angina Unstable (Cardiac disorders) | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 1 | 2
Cardiac Arrest (Cardiac disorders) | 3 | 2
Cardiac Failure (Cardiac disorders) | 2 | 4
Cardiac Failure Acute (Cardiac disorders) | 0 | 2
Cardiac Failure Congestive (Cardiac disorders) | 1 | 3
Cardio-Respiratory Arrest (Cardiac disorders) | 0 | 1
Cardiogenic Shock (Cardiac disorders) | 0 | 1
Coronary Artery Disease (Cardiac disorders) | 0 | 1
Coronary Artery Stenosis (Cardiac disorders) | 1 | 0
Myocardial Infarction (Cardiac disorders) | 1 | 2
Pericardial Effusion (Cardiac disorders) | 0 | 1
Right Ventricular Failure (Cardiac disorders) | 0 | 1
Ventricular Tachycardia (Cardiac disorders) | 0 | 1
Vision Blurred (Eye disorders) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 1
Gastric Haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastric Stenosis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal Angiodysplasia (Gastrointestinal disorders) | 0 | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Impaired Gastric Emptying (Gastrointestinal disorders) | 0 | 1
Inguinal Hernia (Gastrointestinal disorders) | 2 | 2
Intestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Intestinal Obstruction (Gastrointestinal disorders) | 3 | 0
Peptic Ulcer (Gastrointestinal disorders) | 0 | 1
Proctalgia (Gastrointestinal disorders) | 1 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 2
Varices Oesophageal (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 0 | 1
Fatigue (General disorders) | 1 | 0
General Physical Health Deterioration (General disorders) | 1 | 0
Multiple Organ Dysfunction Syndrome (General disorders) | 0 | 1
Non-Cardiac Chest Pain (General disorders) | 1 | 3
Pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 1
Sudden Death (General disorders) | 1 | 3
Biliary Obstruction (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Allergy to Arthropod Sting (Immune system disorders) | 1 | 0
Anaphylactic Reaction (Immune system disorders) | 0 | 1
Alpha Haemolytic Streptococcal Infection (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 0 | 2
Cellulitis (Infections and infestations) | 1 | 1
Clostridium Difficile Infection (Infections and infestations) | 0 | 1
Covid-19 (Infections and infestations) | 1 | 3
Covid-19 Pneumonia (Infections and infestations) | 1 | 2
Cystitis (Infections and infestations) | 0 | 1
Dengue Fever (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Gastroenteritis Salmonella (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 1 | 1
Metapneumovirus Pneumonia (Infections and infestations) | 1 | 0
Necrotising Fasciitis (Infections and infestations) | 1 | 0
Periodontitis (Infections and infestations) | 1 | 0
Pneumocystis Jirovecii Pneumonia (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 10 | 12
Pneumonia Influenzal (Infections and infestations) | 0 | 1
Pneumonia Mycoplasmal (Infections and infestations) | 1 | 0
Pneumonia Respiratory Syncytial Viral (Infections and infestations) | 0 | 1
Psoas Abscess (Infections and infestations) | 1 | 0
Pulmonary Sepsis (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 2
Pyelonephritis Acute (Infections and infestations) | 1 | 0
Respiratory Syncytial Virus Infection (Infections and infestations) | 0 | 1
Respiratory Tract Infection (Infections and infestations) | 0 | 1
Rhinovirus Infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 3 | 5
Septic Shock (Infections and infestations) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 6 | 9
Urosepsis (Infections and infestations) | 3 | 3
Viral Infection (Infections and infestations) | 0 | 1
Ankle Fracture (Injury, poisoning and procedural complications) | 0 | 2
Bladder Injury (Injury, poisoning and procedural complications) | 0 | 1
Cervical Vertebral Fracture (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 4
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 0 | 1
Femur Fracture (Injury, poisoning and procedural complications) | 0 | 3
Fibula Fracture (Injury, poisoning and procedural complications) | 0 | 1
Hand Fracture (Injury, poisoning and procedural complications) | 1 | 1
Head Injury (Injury, poisoning and procedural complications) | 1 | 0
Hip Fracture (Injury, poisoning and procedural complications) | 0 | 2
Joint Injury (Injury, poisoning and procedural complications) | 1 | 0
Multiple Fractures (Injury, poisoning and procedural complications) | 1 | 0
Patella Fracture (Injury, poisoning and procedural complications) | 1 | 0
Procedural Complication (Injury, poisoning and procedural complications) | 1 | 0
Rib Fracture (Injury, poisoning and procedural complications) | 0 | 1
Subdural Haematoma (Injury, poisoning and procedural complications) | 0 | 1
Thermal Burn (Injury, poisoning and procedural complications) | 0 | 1
Tibia Fracture (Injury, poisoning and procedural complications) | 1 | 0
Urinary Tract Stoma Complication (Injury, poisoning and procedural complications) | 0 | 1
Urostomy Complication (Injury, poisoning and procedural complications) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 3
Diabetic Ketosis (Metabolism and nutrition disorders) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 3 | 4
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Chondropathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint Range of Motion Decreased (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 2 | 0
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 4 | 0
Adenocarcinoma Gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastrointestinal Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant Melanoma Stage Iii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Myelodysplastic Syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neuroendocrine Tumour of the Lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ocular Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Papillary Cystadenoma Lymphomatosum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous Cell Carcinoma of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Aphasia (Nervous system disorders) | 0 | 1
Basal Ganglia Infarction (Nervous system disorders) | 1 | 0
Cerebral Artery Occlusion (Nervous system disorders) | 0 | 1
Cerebral Infarction (Nervous system disorders) | 0 | 1
Cerebral Ischaemia (Nervous system disorders) | 1 | 0
Cerebral Venous Sinus Thrombosis (Nervous system disorders) | 1 | 0
Dysarthria (Nervous system disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 1 | 0
Haemorrhagic Stroke (Nervous system disorders) | 0 | 1
Hypoglycaemic Encephalopathy (Nervous system disorders) | 0 | 1
Ischaemic Stroke (Nervous system disorders) | 3 | 2
Memory Impairment (Nervous system disorders) | 0 | 1
Nervous System Disorder (Nervous system disorders) | 0 | 1
Neuralgia (Nervous system disorders) | 0 | 1
Paraparesis (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 0 | 1
Spinal Cord Compression (Nervous system disorders) | 4 | 0
Subarachnoid Haemorrhage (Nervous system disorders) | 1 | 0
Delirium (Psychiatric disorders) | 0 | 1
Disorientation (Psychiatric disorders) | 0 | 1
Mania (Psychiatric disorders) | 0 | 1
Psychotic Disorder (Psychiatric disorders) | 0 | 1
Suicidal Ideation (Psychiatric disorders) | 1 | 0
Acute Kidney Injury (Renal and urinary disorders) | 4 | 6
Bladder Outlet Obstruction (Renal and urinary disorders) | 1 | 0
Bladder Tamponade (Renal and urinary disorders) | 1 | 0
Calculus Bladder (Renal and urinary disorders) | 1 | 1
Calculus Urinary (Renal and urinary disorders) | 1 | 1
Chronic Kidney Disease (Renal and urinary disorders) | 2 | 0
Dysuria (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 5 | 4
Lower Urinary Tract Symptoms (Renal and urinary disorders) | 0 | 1
Ureterolithiasis (Renal and urinary disorders) | 1 | 2
Urethral Stenosis (Renal and urinary disorders) | 0 | 1
Urinary Retention (Renal and urinary disorders) | 3 | 1
Urinary Tract Obstruction (Renal and urinary disorders) | 2 | 2
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Aortic Stenosis (Vascular disorders) | 0 | 1
Essential Hypertension (Vascular disorders) | 0 | 1
Haematoma (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo With Abiraterone Acetate Plus Prednisone (N=348) | Niraparib With Abiraterone Acetate Plus Prednisone (N=347)
Anaemia (Blood and lymphatic system disorders) | 83 | 178
Leukopenia (Blood and lymphatic system disorders) | 18 | 58
Lymphopenia (Blood and lymphatic system disorders) | 26 | 45
Neutropenia (Blood and lymphatic system disorders) | 28 | 74
Thrombocytopenia (Blood and lymphatic system disorders) | 20 | 66
Sinus Tachycardia (Cardiac disorders) | 2 | 21
Abdominal Pain (Gastrointestinal disorders) | 26 | 28
Abdominal Pain Upper (Gastrointestinal disorders) | 14 | 21
Constipation (Gastrointestinal disorders) | 57 | 122
Diarrhoea (Gastrointestinal disorders) | 40 | 51
Dry Mouth (Gastrointestinal disorders) | 14 | 22
Dyspepsia (Gastrointestinal disorders) | 20 | 27
Nausea (Gastrointestinal disorders) | 50 | 107
Vomiting (Gastrointestinal disorders) | 30 | 56
Asthenia (General disorders) | 44 | 47
Fatigue (General disorders) | 64 | 91
Oedema Peripheral (General disorders) | 42 | 55
Pyrexia (General disorders) | 22 | 29
Covid-19 (Infections and infestations) | 70 | 62
Upper Respiratory Tract Infection (Infections and infestations) | 17 | 34
Urinary Tract Infection (Infections and infestations) | 34 | 35
Fall (Injury, poisoning and procedural complications) | 31 | 26
Alanine Aminotransferase Increased (Investigations) | 54 | 22
Aspartate Aminotransferase Increased (Investigations) | 50 | 28
Blood Alkaline Phosphatase Increased (Investigations) | 22 | 14
Blood Creatinine Increased (Investigations) | 16 | 44
Weight Decreased (Investigations) | 18 | 53
Weight Increased (Investigations) | 39 | 12
Decreased Appetite (Metabolism and nutrition disorders) | 18 | 51
Hyperglycaemia (Metabolism and nutrition disorders) | 42 | 48
Hypokalaemia (Metabolism and nutrition disorders) | 69 | 87
Arthralgia (Musculoskeletal and connective tissue disorders) | 74 | 73
Back Pain (Musculoskeletal and connective tissue disorders) | 76 | 66
Bone Pain (Musculoskeletal and connective tissue disorders) | 27 | 18
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 25 | 19
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 39 | 31
Dizziness (Nervous system disorders) | 32 | 50
Headache (Nervous system disorders) | 34 | 47
Insomnia (Psychiatric disorders) | 27 | 49
Dysuria (Renal and urinary disorders) | 21 | 15
Haematuria (Renal and urinary disorders) | 21 | 22
Pollakiuria (Renal and urinary disorders) | 24 | 16
Cough (Respiratory, thoracic and mediastinal disorders) | 40 | 38
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 20 | 45
Hot Flush (Vascular disorders) | 48 | 63
Hypertension (Vascular disorders) | 113 | 152

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2023-08-28): https://cdn.clinicaltrials.gov/large-docs/44/NCT04497844/Prot_000.pdf
  • Statistical Analysis Plan (2025-01-30): https://cdn.clinicaltrials.gov/large-docs/44/NCT04497844/SAP_001.pdf